CLINICAL TRIAL: NCT00691496
Title: A Behavioral Intervention to Reduce Sexual Risk Among African-American Men Who Have Sex With Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centers for Disease Control and Prevention (U.S. Federal Agency)
Collaborators: New York Blood Center (Other); The New York Academy of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CDC-NCHHSTP-5157
Record Dates: First submitted 2008-06-03; First posted 2008-06-05 (Estimated); Last update posted 2012-06-13 (Estimated); Status verified 2012-06

CONDITIONS: HIV Infections
Keywords: HIV Prevention; African-American; gay; bisexual; intervention trial; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Homosexuality; Bisexuality | interventions — Menogaril

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Receives HIV testing and counseling and 5 week intervention
  Interventions: Behavioral: Behavioral intervention to reduce sexual risk among African-American men who have sex with men
- 2 (No Intervention): Receives only HIV Testing and Counseling

INTERVENTIONS:
Behavioral: Behavioral intervention to reduce sexual risk among African-American men who have sex with men — 5 week intervention to increase skill level of participants with talking to their social networks and sexual partners about reducing high risk sexual behaviors while preparing a healthy meal
  Arms: 1

SUMMARY:
The purpose of this project is to test the efficacy of an HIV prevention behavioral intervention to reduce sexual risk among African-American men who have sex with men (MSM).

ELIGIBILITY:
Inclusion Criteria: identify as African-American, Black, Caribbean Black or multiethnic Black, report sex with men

Exclusion Criteria:

* Participated in pilot
* Identify as transgender
* Plan to move before end of study
* Refuse HIV testing at baseline or identified as a newly diagnosed HIV through testing at the baseline
* Under 18 years of age

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 326 (Actual)
Dates: Start 2008-05; Primary Completion 2009-10 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
The primary goal of the intervention is to reduce HIV transmission or acquisition by reducing the frequency of unprotected anal intercourse among African-American MSM. | 3 months after completing intervention

SECONDARY OUTCOMES:
Encourage participants to engage in discussions to reduce sexual risk within their social network and with sexual partners. | 3 months after completing the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Beryl Koblin, PhD, Principal Investigator — New York Blood Center
Locations (1):
- New York Blood Center, New York, New York, United States

REFERENCES:
- [Result] Koblin BA, Bonner S, Powell B, Metralexis P, Egan JE, Patterson J, Xu G, Hoover DR, Goodman K, Chin J, Tieu HV, Spikes P. A randomized trial of a behavioral intervention for black MSM: the DiSH study. AIDS. 2012 Feb 20;26(4):483-8. doi: 10.1097/QAD.0b013e32834f9833. PMID 22156967
- [Result] Tieu HV, Spikes P, Patterson J, Bonner S, Egan JE, Goodman K, Stewart K, Frye V, Xu G, Hoover DR, Koblin BA. Sociodemographic and risk behavior characteristics associated with unprotected sex with women among black men who have sex with men and women in New York City. AIDS Care. 2012;24(9):1111-9. doi: 10.1080/09540121.2012.672723. Epub 2012 Apr 25. PMID 22533637
- [Result] Tieu HV, Xu G, Bonner S, Spikes P, Egan JE, Goodman K, Stewart K, Koblin BA. Sexual partner characteristics, serodiscordant/serostatus unknown unprotected anal intercourse and disclosure among human immunodeficiency virus-infected and uninfected black men who have sex with men in New York City. Sex Transm Dis. 2011 Jun;38(6):548-54. doi: 10.1097/OLQ.0b013e318203e2d7. PMID 21217419